CLINICAL TRIAL: NCT04075344
Title: Effect of a Multimodal Infection Control Program on the Reduction of Bacterial Contamination on Nasogastric Tube Feeding for Elderly Persons in Residential Care Home
Brief Title: Effect of a Infection Control Program on the Reduction of Bacterial Contamination on NG Tube Feeding in RCHEs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ho Suk Ki, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1155074185
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Infection, Bacterial
Keywords: infection control ; bacterial contamination
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Cluster randomized control trials
Who Masked: Outcomes Assessor
Masking Description: This study is single-blinded research, wherein the outcome assessors will be blinded to the assignment of the intervention or control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental RCHEs staff (Experimental): Experimental RCHEs staff will received a multimodal ICP regarding the NG tube feeding. Knowledge and skills of NG tube feeding will be measured before and after the multimodal ICP. In addition, 10 fingertips of RCHEs staff, enteral milk and NG tube hubs of residents will be taken for bacterial counts before and after the intervnetion.
  Interventions: Other: Multimodal Infection control programme
- Control RCHEs staff (No Intervention): No multimodal ICP will be offered to the staff of control RCHEs.

INTERVENTIONS:
Other: Multimodal Infection control programme — 12 weekse educational programme with 6 sessions, 45 minutes per session will be provided to experimental group RCHEs staff
  Arms: Experimental RCHEs staff

SUMMARY:
Septicaemia is a potential complication of nasogastric (NG) tube feeding contamination (Leanne, 2014; Anderton, 2000) and a major cause of morbidity and mortality in residential care home for elders ( RCHEs) (Leanne, 2014). Although health workers (HWs) and personal care workers (PCWs) are responsible for NG tube feeding and direct care to the residents who are fed by NG tube feeding under supervision of registered nurses (RNs) and enrolled nurses (ENs) in RCHEs, HWs and PCWs unfortunately receive limited training regarding infection control (Ho et al., 2012; NICE, 2012; Duckro et al., 2009; Bankhead et al., 2009). A multimodal ICP could reduce the incidence of NG tube feeding contamination by improving the knowledge and skills of RCHE staff members regarding NG tube feeding (Ho et al., 2012). However, because the intervention described by Ho et al. (2012) was not administered in a randomised manner, potential confounders that could affect the outcomes of interest were not adjusted. To overcome that limitation, the proposed work will establish a well-designed multimodal ICP and explore the effectiveness of this intervention in terms of enhancing the knowledge and skills regarding NG tube feeding of RCHE staff members and consequently reducing NG tube feeding contamination after adjusting for potentially important baseline factors.

The proposed research objectives are as follows:

1. To explore the effectiveness of a multimodal ICP for reducing bacterial contamination, as measured by the total bacterial counts on NG tube hubs and fingertips on both hands of RCHEs staff, as well as in enteral milk; and
2. To investigate the effectiveness of a multimodal ICP for improving the knowledge and skills of RCHEs staff members regarding infection control measures during NG tube feeding in RCHEs setting.

DETAILED DESCRIPTION:
In nasogastric tube (NG tube) feeding, a tube is used to transport enteral nutrition to the stomach through the nose (Mosby's Medical Dictionary, 2009). This feeding modality is widely used in the geriatric population, especially for patients with cognitive impairment and oral feeding problems in a residential care home settings (Rowat, 2015). Approximately 3.5% of residents in a Hong Kong residential care home for elders (RCHE) were reported to use NG tubes for long-term feeding (Leung et al., 2000). Contamination of the NG tube hub, defined as the connection port between the NG tube and enteral feeding administration set, is considered a risk factor for the acquisition and transmission of microorganisms (Matlow et al., 2005). NG tube hubs can serve as reservoirs for microorganismal colonisation. For example, enteral milk contamination results from bacterial spread in contaminated tube hubs (Matlow et al., 2005; Donskey, 2004). Accordingly, NG tube feeding contamination occurs when the total bacterial count in enteral milk exceeds 10 to the power 4 colony-forming units per millilitre (cfu/ml) (Borges, Campos, Cardoso, Andre, & Serafini, 2010). NG tube feeding contamination is a serious issue, with potential complications including mortality, septicaemia, bacteraemia, diarrhoea, and pneumonia (Leanne, 2014 & Anderton, 2000).

Previous research indicates that insufficient knowledge about infection control and poor NG tube feeding skills among RCHE staff would result in the passive transport of bacteria from contaminated tube hubs to enteral feed (Ho et al., 2012; National Institute for Health & Clinical Excellence, 2012; Duckro, Blom, Lyle, Weintein, & Hayden, 2009; Bankhead, Boullata, & Brantley, 2009). Additionally, Ho et al. (2012) demonstrated a strong relationship between the number of total bacterial counts on the fingertips of RCHE staff, NG tube hubs of the residents, and enteral milk. In Hong Kong, registered nurses (RNs), enrolled nurses (ENs), health workers (HWs), and personal care workers (PCWs) provide daily nursing care services to residents of RCHEs. Specifically, HWs and PCWs provide direct care, such as NG tube feeding, to residents under the supervision of RNs and ENs. However, PCWs and HWs hold low levels of knowledge and skills related to NG tube feeding (Ho et al., 2012; Annette, Bourgault, Weaver, Swartz, & O'Dea, 2007; Howell, 2002) and receive minimal education on infection control during the care of residents with NG tubes (Hong Kong St. John Ambulance, 2016). Accordingly, the inadequate skills of RCHE staff in terms of NG tube feeding could lead to bacterial contamination (Leanne, 2014; Anderton, 2000).

Despite the above evidence, no previous study has described NG tube feeding practices used at local RCHEs in Hong Kong. Some international studies have revealed that RCHE staff members do not use non-touch techniques when connecting administration sets to the residents' NG tube hubs (Beattie & Anderton, 1998). Annette et al. (2007) reported that RCHE staff members unnecessarily disconnected NG tube feeding systems while repositioning residents and changing linens. Moreover, although 60-ml syringes are widely recommended for the prevention of multi-decanting procedures when administrating milk and medications (Roberts et al., 2007; Bowers, 2000), a previous study found that RCHE staff members repeatedly used 20-ml syringes during milk and medication decanting procedures (Annette et al., 2007). NICE (2012) advised the use of sterile water to flush all feeding tubes. However, in one study, RCHE staff used non-boiled water during NG tube feeding in elderly residents (Allen, 2015). These poor skills increase the risk of bacterial growth in NG tube feeding systems (NICE, 2012 & Ho et al., 2102).

A previous study reported a relationship among NG tube hub contamination, NG tube feeding contamination, and insufficient NG tube feeding knowledge and skills held by RCHE staff members (Ho et al., 2012). Therefore, a comprehensive literature search was conducted to explore the effects of an infection control education programme on NG tube feeding contamination in RCHEs. Four studies conducted at RCHEs in the United States (Michigan), Europe (Northern Ireland and France) and Hong Kong satisfied the literature search objectives (Mody, Krein, Saint, Min, Montoya & Lansing, 2015; Ho et al., 2012; Kathleen, Gavazzi, Bar-Hen, Carrat, de Wazieres, & Lejeune, 2012; Baldwin, Gilpin, Tunney, Kearney, Crymble, & Cardwell, 2010). These four studies featured several common characteristics of teaching contents, including the provision of a multimodal infection control programme (ICP) regarding hand hygiene education, the proper use of personal protective equipment, and medical device (NG tube) care to RCHE staff. The studies utilised a combination of multimodal strategies with varied multimodal ICP contents. Here, 'multimodal' is defined as the involvement of several modes of activities, whereas 'strategy' is defined as a plan of action intended to accomplish a specific goal (Free Dictionary Oxford, 2016). Therefore, a multimodal strategy is needed to improve infection control practice (Pittet et al., 2000).

The proposed multimodal ICP will have a duration of 12 weeks to ensure the sustainability of knowledge and skills. Six 45-minute sessions will be provided at 2-week intervals.

In this study, the investigator would explore the effectiveness of the multimodal ICP in the reduction of the total bacterial counts on the NG tube hubs, enteral millk of the residents and the 10 fingertips of the RCHEs staff by increasing the knowledge and skills of the NG tube feeding among RCHEs staff with the multimodal ICP.

ELIGIBILITY:
Inclusion criteria of RCHEs:

The investigator will search the Hong Kong Social Welfare Department website to determine which RCHEs should be invited based on the following inclusion criteria:

1. Chinese facilities licensed under The Hong Kong Social Welfare Department;
2. provision of NG tube feeding service to elders;
3. provision of nursing care services to elders by RNs, ENs, HWs, and PCW;
4. government subsidisation [either subvented homes operated by non-government organisations (NGOs) or private homes participating in an Enhanced Bought Place Scheme (EBPS), EA1]; and
5. consent to participate and assurance that the entire staff team will join the study.

Exclusion criteria of RCHEs:

1. RCHEs do not provide NG tube feeding to residents.
2. RCHEs do not assurance the entire staff team will join the study.

Inclusion Criteria of Residential care home staff: :

1. RCHEs staff members (RNs, ENs, HWs, and PCWs) who participate in the daily care of residents at the selected RCHEs.
2. RCHEs staff can read Chinese and speak Cantonese.

Exclusion criteria of Residential care home staff::

1. RCHEs staff do not understand Chinese
2. RCHEs staff do not participate in NG tube feeding

Inclusion criteria of residents:

(1) All residents receiving NG tube feeding in the participating homes will be included.

Exclusion Criteria of residents:

1. Residents in whom NG tube feeding is assisted by relatives or caregivers other than RCHE staff members.
2. Residents with presence of transmission-based precautions, such as airborne, contact, or droplet contamination will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2019-09-02 (Estimated); Primary Completion 2020-04-29 (Estimated); Study Completion 2020-04-29 (Estimated)

PRIMARY OUTCOMES:
A change of total bacterial counts on NG tube hubs | Before and after the intervention (4 months aparts)
  A sampling will be taken to the residents' NG tube hubs for the measuring the total bacterial counts (cfu/ml) to investigate if there will have any changes after 4 months.
  NG tube feeding contamination occurs when the total bacterial count in enteral milk exceeds10 to the power 4 colony-forming units per millilitre (cfu/ml) (Borges, Campos, Cardoso, Andre, & Serafini, 2010). Therefore total bacterial counts of NG tube hubs exceed 10 to the power 4 cfu/ml is considered contamination.

SECONDARY OUTCOMES:
A change of total bacterial counts on enteral milk of residents | Before and after the intervention (4 months aparts)
  A sampling will be taken to the enteral milk of residents for the measuring the total bacterial counts (cfu/ml) to investigate if there will have any changes after 4 months.
  Total bacterial counts of enteral milk exceeds 10 to the power 4 cfu/ml is considered contamination.
A change of skills on the NG tube feeding among the RCHEs staff | Before and after the intervention (4 months aparts)
  RCHEs staff 's skills on NG tube feeding will be assessed by outcomes assessors to investigate if there will have any changes after 4 months.
  Investigator will use "Skill Assessment form regarding NG tube feeding" which was developed by Ho et al. (2012). This form comprises 32 items regarding NG tube feeding procedure. One point will be awarded for each requirement achieved by the RCHE staff member. The total maximum score is 32 points, and a higher score indicates better NG tube feeding skills. The content validity of this assessment is 0.86, and the test-retest reliability is 0.82.
A change of Knowledge on the NG tube feeding among the RCHEs staff | Before and after the intervention (4 months aparts)
  RCHEs staff will be required to complete the knowledge questionnaire regarding the NG tube feeding to investigate if there will have any changes after 4 months.
  The investigator will use "self-administered questionnaire regarding knowledge about NG tube feeding" which was developed by Ho et al. (2012). This questionnaire comprises 20 true/false items, and each correct answer is given one point. The total maximum score is 20 points, and a higher score indicates better knowledge in the area of infection control related to NG tube feeding. The content validity index of this questionnaire is 1.0, and the test-retest reliabilty is 0.84.
A change of total bacterial counts on 10 fingertips of RCHEs staff | Before and after the intervention (4 months aparts)
  A sampling will be taken to the 10 fingertips of RCHEs staff for the measuring the total bacterial counts (cfu/ml) to investigate if there will have any changes after 4 months.
  Total bacterial counts of 10 fingertips exceed 10 to the power 4 cfu/ml is considered contamination.

CONTACTS AND LOCATIONS:
Overall Officials: Suki Ho, Msc, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baldwin NS, Gilpin DF, Tunney MM, Kearney MP, Crymble L, Cardwell C, Hughes CM. Cluster randomised controlled trial of an infection control education and training intervention programme focusing on meticillin-resistant Staphylococcus aureus in nursing homes for older people. J Hosp Infect. 2010 Sep;76(1):36-41. doi: 10.1016/j.jhin.2010.03.006. Epub 2010 May 7. PMID 20451294
- [Background] Chami K, Gavazzi G, Bar-Hen A, Carrat F, de Wazieres B, Lejeune B, Armand N, Rainfray M, Hajjar J, Piette F, Rothan Tondeur M. A short-term, multicomponent infection control program in nursing homes: a cluster randomized controlled trial. J Am Med Dir Assoc. 2012 Jul;13(6):569.e9-17. doi: 10.1016/j.jamda.2012.04.008. Epub 2012 Jun 7. PMID 22682697
- [Background] Mody L, Krein SL, Saint S, Min LC, Montoya A, Lansing B, McNamara SE, Symons K, Fisch J, Koo E, Rye RA, Galecki A, Kabeto MU, Fitzgerald JT, Olmsted RN, Kauffman CA, Bradley SF. A targeted infection prevention intervention in nursing home residents with indwelling devices: a randomized clinical trial. JAMA Intern Med. 2015 May;175(5):714-23. doi: 10.1001/jamainternmed.2015.132. PMID 25775048
- [Result] Ho SS, Tse MM, Boost MV. Effect of an infection control programme on bacterial contamination of enteral feed in nursing homes. J Hosp Infect. 2012 Sep;82(1):49-55. doi: 10.1016/j.jhin.2012.05.002. Epub 2012 Jul 4. PMID 22765960